CLINICAL TRIAL: NCT02149615
Title: Prospective Open-label Phase IV Trial to Investigate the Frequency of Optic Disc Swelling, Idiopathic Intracranial Hypertension and Dry Eye Symptoms Under Antiacne Medication Treatment
Brief Title: Antiacne Medications Pseudotumor Cerebri
Acronym: AAMPTC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH 2013-0433 AAMPTC; 2013DR4066 (Other: Swiss Medic)
Record Dates: First submitted 2014-04-07; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Optic Disc Swelling
Keywords: idiopathic intracranial hypertension; optic disc swelling; antiacne medication; isotretinoin
MeSH Terms: conditions — Papilledema; Pseudotumor Cerebri

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- isotretinoin (Experimental): Retinal nerve fibre layer measurement in patients under isotretinoin treatment
  Interventions: Other: Retinal nerve fibre layer measurement
- lymecycline (Active Comparator): Retinal nerve fibre layer measurement in patients under lymecycline treatment
  Interventions: Other: Retinal nerve fibre layer measurement
- minocycline (Active Comparator): Retinal nerve fibre layer measurement in patients under minocycline treatment
  Interventions: Other: Retinal nerve fibre layer measurement
- doxycycline (Active Comparator): Retinal nerve fibre layer measurement in patients under doxycycline treatment
  Interventions: Other: Retinal nerve fibre layer measurement

INTERVENTIONS:
Other: Retinal nerve fibre layer measurement — Measurement of retinal nerve fibre layer thickness using optic coherence tomography.
  Other Names: effect of medication on optic nerve fibre layer

SUMMARY:
The exact incidence of optic disc swelling and idiopathic intracranial hypertension in patients using antiacne medication is not known so far. The investigators hypothesize that swelling of retinal nerve fibre layer measured by optical coherence tomography is more frequent then assumed so far.

DETAILED DESCRIPTION:
Measurement of retinal nerve fibre layer using optical coherence tomography over a period of 6 to 9 months depending on exact antiacne medication.

ELIGIBILITY:
Inclusion Criteria:

* Antiacne medication treatment indicated by dermatologist
* age > 18 years
* contraception if indicated

Exclusion Criteria:

- age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fibre layer | 9 months
  Measurement of retinal nerve fibre layer using optical coherence tomography. Changes over 10 micrometers are considered to be clinically relevant.
  The Term "retinal nerve fibre layer" describes an automated standardized optical coherence tomography measurement program measuring the sectorial thickness of the peripapillar retinal nerve fibre layer. There exists no other term for that.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Landau, Prof MD, Study Chair — UniversityHospital, Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- See also: Study register Switzerland — http://www.kofam.ch